CLINICAL TRIAL: NCT04337918
Title: Multi-Center, Randomized, Controlled, Phase II Clinical Efficacy Study Evaluating Nitric Oxide Releasing Solution Treatment for the Prevention and Treatment of COVID-19 in Healthcare Workers and Individuals at Risk of Infection
Brief Title: Nitric Oxide Releasing Solutions to Prevent and Treat Mild/Moderate COVID-19 Infection
Acronym: NOCOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Collaborators: The Emmes Company, LLC (Industry); Keyrus Life Science (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COVID-CTP-01
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Corona Virus Infection
Keywords: Antiviral; Virucidal; Nitric Oxide
MeSH Terms: conditions — Coronavirus Infections | interventions — noggin protein

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized, controlled, phase II, parallel group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prevention - Standard Precautions (No Intervention): Participants COVID-19 negative at baseline will be randomized to receive standard COVID-19 screening and protection (per their facility or organization's protocols).
- Prevention - NORS + Standard Precautions (Experimental): Participants COVID-19 negative at baseline will be randomized to receive standard COVID-19 screening and protection (per their facility or organization's protocols) plus daily NORS treatment for 14 days.
  Interventions: Drug: NORS (Nitric Oxide Releasing Solution)
- Treatment Sub-Study (Other): Volunteers who are found to be COVID-19 positive during screening will be eligible to enroll in the 21-day Treatment sub-study and receive daily NORS treatment for 14 days. Ten participants can be directly enrolled in the Treatment sub-study.
  Participants enrolled in the Prevention study who meet the criteria in this section will roll over into the Treatment Sub-Study but must remain in their randomly assigned group.
  Interventions: Drug: NORS (Nitric Oxide Releasing Solution)

INTERVENTIONS:
Drug: NORS (Nitric Oxide Releasing Solution) — NORS treatment will consist of daily self-administration of three routes; Nitric Oxide Gargle (NOG) every morning, Nitric Oxide Nasophyaryngeal Irrigation (NONI) every evening, and Nitric Oxide Nasal Spray (NONS) up to 5 times per day.
  Other Names: NOG, NONI, NONS
  Arms: Prevention - NORS + Standard Precautions
Drug: NORS (Nitric Oxide Releasing Solution) — Up to ten volunteers who are found to be COVID-19 positive during screening will be eligible to enroll in the 21-day Treatment sub-study and receive daily NORS treatment for 14 days. NORS treatment will consist of daily self-administration of three routes; Nitric Oxide Gargle (NOG) every morning, Nitric Oxide Nasophyaryngeal Irrigation (NONI) every evening, and Nitric Oxide Nasal Spray (NONS) up to 5 times per day.
  Any participants enrolled in the Prevention study who meet the criteria for the sub study will roll over into the Treatment Sub-Study but must remain in their randomly assigned group.
  Other Names: NOG, NONI, NONS
  Arms: Treatment Sub-Study

SUMMARY:
This is a multi-center, randomized, controlled, phase II clinical efficacy study evaluating a novel Nitric Oxide Releasing Solution (NORS) treatment for the prevention and treatment of COVID-19 in healthcare workers at risk of infection. Participants will be enrolled into one of two components of this study. Based on initial swabs/symptoms, volunteers who are COVID-19 negative will be enrolled in the Prevention study and randomized to receive standard institutional precautions or standard institutional precautions + NORS. Those who are COVID-19 positive will be enrolled in the open-label Treatment Sub-Study.

DETAILED DESCRIPTION:
The novel, human-infecting corona-virus, provisionally named 2019 novel corona virus (2019-nCoV) is a single-strand, positive-sense RNA virus and has a similar receptor-binding domain structure to that of SARS-CoV and MERS-CoV. The virus is transmitted via airborne droplets to the nasal mucosa. Replication occurs locally in the nasal mucosa, in ciliated epithelial cells, over a 3-day incubation period. The mucosal cells are damaged with a resultant inflammatory response similar to the common cold. During this time the virus is shed in nasal secretions causing disease in the lower respiratory tract, potentially causing fatal viral pneumonia.

The literature supports that NO or its derivatives have inhibitory effects on a variety of viral infections. This inhibitory effect was shown to be marked in Interferon (IFN) mediated inhibition manifested by activated macrophage. It was also shown to be correlated with s-nitrosylation of viral proteins such as reductases and proteases.

Based on the genetic similarities between SARS and corona viruses, similar viricidal effects of NO on COVID-19 can be hypothesized.

SaNOtize has developed an innovative approach to provide nitric oxide gas using a formulation called Nitric Oxide Releasing Solution (NORS). This patented solution releases virucidal doses of NO for a sustained period and is effective at rapidly inactivating Influenza A and SARS-CoV-2.

NORS delivered as a gargle (AM), nasal spray (PRN) or as a nasopharyngeal flush (PM) has the potential to decontaminate the upper respiratory tract that could preventing transmission and progression of COVID-19 in Healthcare Workers & Individuals at Risk of Infection.

The randomized Prevention study will investigate the ability of NORS to prevent COVID-19 infection when used prophylactically. The open-label Treatment Sub-Study is expected to be small and will provide pilot data on the possibility of NORS as a treatment for Mild/Moderate COVID-19 infection.

ELIGIBILITY:
Prevention Study Inclusion Criteria:

1. Capable of understanding and providing signed informed consent and ability to adhere to the requirements and restrictions of this protocol;
2. Men and Women ≥ 19 years of age unless local laws dictate otherwise;
3. English speaking;
4. Must be willing to use an adequate form of contraception (or abstinence) from the time of the first dose with the IMP until after the last dose of IMP.
5. Be symptom-free at screening/baseline.
6. Work/live in contact with COVID-19 infected patients or scheduled to work in a setting with high likelihood of contact with COVID-19 infected patients.

Prevention Study Exclusion Criteria:

1. Prior Tracheostomy;
2. Concomitant treatment of respiratory support (involving any form of oxygen therapy);
3. Any clinical contraindications, as judged by the attending physician;
4. Any symptoms consistent with COVID-19;
5. Pregnant;
6. Mentally or neurologically disabled patients who are considered not fit to consent to their participation in the study;
7. Prior COVID-19 infection.

Treatment Sub study Inclusion Criteria:

1. Capable of understanding and providing signed informed consent and ability to adhere to the requirements and restrictions of this protocol;
2. Men and Women ≥ 19 years of age unless local laws dictate otherwise;
3. English speaking;
4. Must be willing to use an adequate form of contraception (or abstinence) from the time of the first dose with the IMP until after the last dose of IMP;
5. Positive COVID-19 test or presentation of clinical symptoms defined as fatigue with either fever >37.2 (oral) and/or a persistent cough.

Treatment Sub Study Exclusion Criteria:

1. Prior Tracheostomy;
2. Concomitant treatment of respiratory support (involving any form of oxygen therapy); Any clinical contraindications, as judged by the attending physician;
3. Mentally or neurologically disabled patients who are considered not fit to consent to their participation in the study;
4. Pregnant;
5. Currently hospitalized for symptoms of COVID-19.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Prevention Study: Measure the effect of NORS on the prevention of COVID-19 infection among health care professionals at risk of exposure to COVID-19 | 14 days
  Measure the proportion of subjects with either swab positive COVID-19 or presentation of clinical symptoms as measured by fatigue with either fever >37.2 (oral)and/or a persistent cough.
Treatment Sub Study: Measure the efficacy of NORS at reducing the progression of COVID- 19 | 21 days
  Measure the proportion of participants requiring requiring hospitalization for COVID-19/flu-like symptoms and/or needing oxygen therapy, BIPAP/CPAP, intubation and mechanical ventilation following enrollment.

SECONDARY OUTCOMES:
Prevention Study: Measure the effect of NORS on the prevention of progression of COVID- 19 | 21 days
  Measure the proportion of participants requiring requiring hospitalization for COVID-19/flu-like symptoms and/or needing oxygen therapy, BIPAP/CPAP, intubation and mechanical ventilation following enrollment.
Prevention Study: Measure the tolerability of NORS treatments | 21 days
  Measure the tolerability of the NORS treatments as determined by number of adverse events, pain, discomfort or discontinuations of treatment.
Treatment Sub Study: Measure the virucidal effect of NORS Treatments | 21 days
  Measure the median number of days to negative conversion of SARS-CoV-2 RT-PCR from a nasopharyngeal swabs.
Treatment Sub Study: Determine effect of NORS on the speed of clinical recovery | 21 days
  Determine the time to clinical recovery in participants with COVID-19 by measuring the median number of days from enrollment to discharge (if admitted), or to normalization of fever (defined as <36.6°C from axillary site, or < 37.2°C from oral site or < 37.8°C from rectal or tympanic site), respiratory rate (< 24 bpm while breathing room air).
Treatment Sub Study: Determine the reduction in clinical symptoms | 21 days
  Measure the reduction clinical symptoms in participants with COVID- 19 by the magnitude of the change in Modified Jackson Cold Score Diary Score (5-unit change is a substantial clinical benefit).
Treatment & Sub Study: Determine positive sero-conversion for SARS-CoV-2 | 21 days
  Measure the proportion of participants that have a positive sero-conversion for SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Road, MD, Principal Investigator — Private Practice
Locations (5):
- Canada (5):
  - BC Diabetes, Vancouver, British Columbia
  - LMC Manna, Pointe-Claire, Quebec
  - Diex Recherche Québec, Québec, Quebec
  - Diex Recherche Joliette, Saint-Charles-Borromée, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reiss CS, Komatsu T. Does nitric oxide play a critical role in viral infections? J Virol. 1998 Jun;72(6):4547-51. doi: 10.1128/JVI.72.6.4547-4551.1998. No abstract available. PMID 9573217
- [Background] Colasanti M, Persichini T, Venturini G, Ascenzi P. S-nitrosylation of viral proteins: molecular bases for antiviral effect of nitric oxide. IUBMB Life. 1999 Jul;48(1):25-31. doi: 10.1080/713803459. PMID 10791912
- [Background] Deppisch C, Herrmann G, Graepler-Mainka U, Wirtz H, Heyder S, Engel C, Marschal M, Miller CC, Riethmuller J. Gaseous nitric oxide to treat antibiotic resistant bacterial and fungal lung infections in patients with cystic fibrosis: a phase I clinical study. Infection. 2016 Aug;44(4):513-20. doi: 10.1007/s15010-016-0879-x. Epub 2016 Feb 9. PMID 26861246
- [Background] Miller CC, Hergott CA, Rohan M, Arsenault-Mehta K, Doring G, Mehta S. Inhaled nitric oxide decreases the bacterial load in a rat model of Pseudomonas aeruginosa pneumonia. J Cyst Fibros. 2013 Dec;12(6):817-20. doi: 10.1016/j.jcf.2013.01.008. Epub 2013 Mar 6. PMID 23481089
- [Background] Miller C, Miller M, McMullin B, Regev G, Serghides L, Kain K, Road J, Av-Gay Y. A phase I clinical study of inhaled nitric oxide in healthy adults. J Cyst Fibros. 2012 Jul;11(4):324-31. doi: 10.1016/j.jcf.2012.01.003. Epub 2012 Apr 18. PMID 22520076
- [Background] McMullin BB, Chittock DR, Roscoe DL, Garcha H, Wang L, Miller CC. The antimicrobial effect of nitric oxide on the bacteria that cause nosocomial pneumonia in mechanically ventilated patients in the intensive care unit. Respir Care. 2005 Nov;50(11):1451-6. PMID 16253152
- [Background] Regev-Shoshani G, Vimalanathan S, McMullin B, Road J, Av-Gay Y, Miller C. Gaseous nitric oxide reduces influenza infectivity in vitro. Nitric Oxide. 2013 May 31;31:48-53. doi: 10.1016/j.niox.2013.03.007. Epub 2013 Apr 2. PMID 23562771
- [Background] Regev-Shoshani G, McMullin B, Nation N, Church JS, Dorin C, Miller C. Non-inferiority of nitric oxide releasing intranasal spray compared to sub-therapeutic antibiotics to reduce incidence of undifferentiated fever and bovine respiratory disease complex in low to moderate risk beef cattle arriving at a commercial feedlot. Prev Vet Med. 2017 Mar 1;138:162-169. doi: 10.1016/j.prevetmed.2015.04.008. Epub 2015 Apr 20. PMID 25975664